CLINICAL TRIAL: NCT02860910
Title: Cross-Cultural Cognitive Behavioral Group Therapy: Evaluating the Effectiveness of a Manualized Cognitive Behavior Group Therapy Treatment for the Management of Menopause Symptoms in a Mood and Anxiety Disorder Population
Brief Title: Cognitive Behavioral Group Therapy for the Management of Menopause Symptoms in Mood Disorders
Acronym: Conklin MWW
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Danette Conklin, PhD (Other)
Responsible Party: Sponsor-Investigator, Danette Conklin, PhD, Director of Midlife Wellness for Woman, University Hospitals Cleveland Medical Center
Organization: University Hospitals Cleveland Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 04-16-11
Record Dates: First submitted 2016-06-14; First posted 2016-08-09 (Estimated); Last update posted 2019-09-30 (Actual); Status verified 2019-09

CONDITIONS: Bipolar Disorder; Major Depressive Disorder; Menopause
Keywords: hot flashes; postmenopause; perimenopause
MeSH Terms: conditions — Bipolar Disorder; Depressive Disorder, Major; Hot Flashes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Cognitive Behavioral Group Therapy (Experimental): The six CBGT sessions are outlined in the manual entitled: Managing Hot Flushes with Group Cognitive Behaviour Therapy: An Evidenced-Based Treatment Manual for Health Care Professionals (Hunter & Smith, 2015) as follows:
  Session 1: Psycho-education and the cognitive behavioural model Session 2: Stress management, improving wellbeing and identifying precipitants Session 3: Managing hot flushes using a cognitive behavioural approach Session 4: Managing night sweats and improving sleep (part one) Session 5: Managing night sweats and improving sleep (part two) Session 6: Review and maintaining changes (One alteration: Open discussion about mood disorders, anxiety and the psychological impact instead of the psychological impact of breast cancer)
  Interventions: Behavioral: Cognitive Behavioral Group Therapy

INTERVENTIONS:
Behavioral: Cognitive Behavioral Group Therapy

SUMMARY:
The general objective of this study is to advance insight into non-pharmacological treatments for maturing women that impact psychological health and wellbeing of women adapting to menopause, a natural but often challenging developmental milestone.

DETAILED DESCRIPTION:
This exploratory study proposes to expand the knowledge in the menopausal literature and evaluate the effectiveness of cognitive-behavioral group therapy (CBGT) in reducing problematic vasomotor symptoms, reducing daily interference and improving quality of life. The study will include two homogenous peri- or post-menopausal cohorts (African-American and Caucasian) with major depressive disorder or bipolar disorder. The intervention will be delivered in groups of 6 to 10 participants per group of both race/ethnicities in an outpatient setting during a 6-week time period. The participants will be assessed on the degree of hot flash problem rating, hot flash related daily interference, and menopause quality of life at screening, baseline, and post-treatment. Participants will also be assessed using the following predictor variables at the same time points: body mass index (BMI), level of perceived stress, severity of depression, severity of anxiety level of pleasure, severity of mania, hot flash beliefs and severity of couple's conflict.

ELIGIBILITY:
Inclusion Criteria.

1. Self-identified as African-American or Caucasian females between 40-65 experiencing the early, late peri-menopause or early or late post-menopause stages of reproductive aging defined by The North American Menopause Society (NAMS, 2014), Menopause Practice guidelines, stages of reproductive aging. There are situations in which menopause status will not be able to be determined, such as with women who have had a hysterectomy. However, if the potential study participant meets all other inclusion criteria, then she can be enrolled in the study.
2. Diagnosed with current or lifetime bipolar disorder or major depressive disorder as assessed by the MINI International Neuropsychiatric Interview (MINI) for Diagnostic and Statistical Manual-5 (DSM-5).
3. Menopause symptoms can be natural or surgically induced.
4. Willing to remain on current dose of psychotropic medications until the study has concluded.
5. Experiencing one or more hot flashes and/or night sweats per day.
6. Willing to have the 6 CBGT interventions audio recorded.
7. English speaking with at least a high school education.
8. Montgomery-Asberg Depression Rating Scale (MADRS) total score > 7
9. Women stable on psychotropic medications for ≥ 8 weeks.

Medication regimens to treat their DSM-V diagnoses will be encouraged to continue in order to determine if the CBGT accounted for any change in symptoms.

Exclusion Criteria.

1. Unwilling or unable to comply to study requirements.
2. Women diagnosed with schizophrenia, schizoaffective, borderline personality disorder, and/or active psychosis, as confirmed by MINI.
3. Diagnosed with active substance use disorder within past 12 months as confirmed on the MINI.
4. Women currently treated with hormone therapy (HT) for Vasomotor Symptoms (VMS).
5. Diagnosed with current post-traumatic stress disorder (PTSD).
6. Participants experiencing acute mania as defined by a Young Mania Rating Scale (YMRS) score > 15
7. Serious suicidal risks judged by the investigator or having score equal or greater than 4 on MADRS item number 10 at screening or baseline.
8. Participants being treated with chemotherapy and/or tamoxifen.
9. Women who are not self-identifying as either African-American or Caucasian.

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2018-10 (Actual); Study Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
Number of participants who begin cognitive group behavioral therapy | 2 years
Change in Hot Flush Rating Scale: Frequency and Problem Rating (HFRS) total score | Baseline and Week 6

SECONDARY OUTCOMES:
Change in Hot Flash Daily Interference Scale (HFRDIS) total score | Baseline and Week 6
Change in Menopause Representation Questionnaire (MRQ) total score | Baseline and Week 6

CONTACTS AND LOCATIONS:
Overall Officials: Danette Conklin, PhD, Principal Investigator — University Hospitals Cleveland Medical Center
Locations (1):
- University Hospitals Cleveland Medical Center - Mood Disorders Program, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Conklin D, Carpenter JS, Whitney MS, DeLozier S, Ogede DO, Bazella C, McVoy M, Sajatovic M. Narrative Analyses: Cognitive Behavior Group Therapy for Women with Menopause and Bipolar or Major Depressive Disorders. Womens Health Rep (New Rochelle). 2021 Sep 22;2(1):430-442. doi: 10.1089/whr.2021.0025. eCollection 2021. PMID 34671764
- [Derived] Conklin DY, Goto T, Ganocy S, Loue S, LaGrotta C, Delozier S, Brownrigg B, Conroy C, D'Arcangelo N, Janes J, Ogede D, Sajatovic M. Manualized cognitive behavioral group therapy to treat vasomotor symptoms for women diagnosed with mood disorders. J Psychosom Res. 2020 Jan;128:109882. doi: 10.1016/j.jpsychores.2019.109882. Epub 2019 Nov 20. PMID 31837624

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-04-18): https://cdn.clinicaltrials.gov/large-docs/10/NCT02860910/Prot_SAP_000.pdf